CLINICAL TRIAL: NCT05753423
Title: Impact of Maternal Depression, Anxiety, Stress, and Perceived Social Support on the Oral Health Status and Oral Health-related Quality of Life of Their Children
Brief Title: Impact of Maternal Mental Health on the Oral Health Status and Oral Health-related Quality of Life of Their Children
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Yehia, Assistant Lecturer at Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University
Other Study IDs: DPH 22-1D
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Disorder; Oral Health-Related Quality of Life
Keywords: Mental Health; Social support; Oral Health-Related Quality of Life
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian mothers-children pairs: Egyptian mothers-children pairs attending the Faculty of Dentistry, Ain Shams University will be recruited.
  Interventions: Diagnostic Test: Interview-based questionnaires & Clinical examination

INTERVENTIONS:
Diagnostic Test: Interview-based questionnaires & Clinical examination — Interview-based questionnaires will be conducted among Egyptian mothers attending Pediatric Dentistry and Dental Public Health outpatient clinic at Faculty of Dentistry, Ain Shams University by the principal investigator. Clinical examination of the oral health status of their preschool children aged 3-5 years will be conducted by the principal investigator.

SUMMARY:
Dental caries is a complex multifactorial disease that is strongly related to and influenced by the children's dietary habits, sugar intake, salivary flow, salivary fluoride level, and preventive behaviors. Based on the literature, other factors can affect child dental caries including the influence of social factors, such as the family environment. To avoid suffering from dental caries, preventive oral hygiene practices beginning in childhood are crucial. However, parents are the primary providers of oral health care for their children and they generally play a pivotal role in the overall health and oral health of both children and adolescents. Therefore, this study aims to investigate the impact of maternal mental health in the form of depression, anxiety, or stress and their perceived social support on the oral health status and OHRQoL of their children.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian mothers.
* Preschool children of both sexes aged (3-5 years who have a full set of primary dentition).
* Healthy children with no long-term medications, and with no physical, learning, or mental disabilities.

Exclusion Criteria:

* Mothers who do not consent to participate in the study (either for themselves or for their children)
* Mothers with any diagnosed mental disorders.
* Pregnant mothers or mothers who delivered within the last year.
* Mothers with any diagnosed physical disabilities.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian mothers-children pairs: preschool children of both sexes aged 3-5 years who have a full set of primary dentition and their mothers.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
The presence of maternal mental issue in the form of depression, anxiety, or stress | 1 year
  The mental health of Egyptian mothers is assessed through the validated Arabic form of the depression anxiety stress scale-21 (DASS-21).
The caries experience of their children (aged 3-5 years) | 1 year
  Dental caries experience is estimated by calculating the three components (decayed, missed, and filled) of the dmft index for primary teeth according to World Health Organization (WHO).
The oral hygiene status of their children (aged 3-5 years) | 1 year
  Oral hygiene is assessed by the debris component of the modified form of Oral Hygiene Index-Simplified (OHI-S) that can be used for deciduous teeth.
Oral health-related quality of life of their children | 1 year
  A validated Arabic version of the Early Childhood Oral Health Impact Scale (ECOHIS) is used to examine mothers' perceptions of their preschool children's oral health-related quality of life (OHRQoL).

SECONDARY OUTCOMES:
The perceived social support of Egyptian mothers | 1 year
  The perceived social support of Egyptian mothers is assessed by the multidimensional scale of perceived social support (Arabic- MSPSS).
The oral health-related behaviors of their children | 1 year
  Egyptian mothers are asked five questions about their children's snacking habit, frequency of tooth brushing, brushing with or without adult assistance, and dental visit utilization and pattern. These questions were adopted from previous similar studies in English and then were translated into Arabic.
The perception of Egyptian mothers about the dental health status of their children | 1 year
  Participants are asked to rate the dental health status of their children on a 5-point scale from 'very good' to 'very poor'.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Oral Disorders Collaborators; Bernabe E, Marcenes W, Hernandez CR, Bailey J, Abreu LG, Alipour V, Amini S, Arabloo J, Arefi Z, Arora A, Ayanore MA, Barnighausen TW, Bijani A, Cho DY, Chu DT, Crowe CS, Demoz GT, Demsie DG, Dibaji Forooshani ZS, Du M, El Tantawi M, Fischer F, Folayan MO, Futran ND, Geramo YCD, Haj-Mirzaian A, Hariyani N, Hasanzadeh A, Hassanipour S, Hay SI, Hole MK, Hostiuc S, Ilic MD, James SL, Kalhor R, Kemmer L, Keramati M, Khader YS, Kisa S, Kisa A, Koyanagi A, Lalloo R, Le Nguyen Q, London SD, Manohar ND, Massenburg BB, Mathur MR, Meles HG, Mestrovic T, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mokdad AH, Morrison SD, Nazari J, Nguyen TH, Nguyen CT, Nixon MR, Olagunju TO, Pakshir K, Pathak M, Rabiee N, Rafiei A, Ramezanzadeh K, Rios-Blancas MJ, Roro EM, Sabour S, Samy AM, Sawhney M, Schwendicke F, Shaahmadi F, Shaikh MA, Stein C, Tovani-Palone MR, Tran BX, Unnikrishnan B, Vu GT, Vukovic A, Warouw TSS, Zaidi Z, Zhang ZJ, Kassebaum NJ. Global, Regional, and National Levels and Trends in Burden of Oral Conditions from 1990 to 2017: A Systematic Analysis for the Global Burden of Disease 2017 Study. J Dent Res. 2020 Apr;99(4):362-373. doi: 10.1177/0022034520908533. Epub 2020 Mar 2. PMID 32122215
- [Background] Lorber MF, Maisson DJ, Slep AM, Heyman RE, Wolff MS. Mechanisms Linking Interparental Aggression to Child Dental Caries. Caries Res. 2017;51(2):149-159. doi: 10.1159/000453672. Epub 2017 Jan 28. PMID 28132053
- [Background] Alshammari FS, Alshammari RA, Alshammari MH, Alshammari MF, Alibrahim AK, Al Sineedi FA, Alkurdi KA, Alshammari AF. Parental Awareness and Knowledge toward their Children's Oral Health in the City of Dammam, Saudi Arabia. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):100-103. doi: 10.5005/jp-journals-10005-1894. PMID 34326593
- [Background] Abanto J, Carvalho TS, Mendes FM, Wanderley MT, Bonecker M, Raggio DP. Impact of oral diseases and disorders on oral health-related quality of life of preschool children. Community Dent Oral Epidemiol. 2011 Apr;39(2):105-14. doi: 10.1111/j.1600-0528.2010.00580.x. Epub 2010 Oct 5. PMID 21029148
- [Background] Alkan A, Cakmak O, Yilmaz S, Cebi T, Gurgan C. Relationship Between Psychological Factors and Oral Health Status and Behaviours. Oral Health Prev Dent. 2015;13(4):331-9. doi: 10.3290/j.ohpd.a32679. PMID 25197739
- [Background] Costa FDS, Azevedo MS, Ardenghi TM, Pinheiro RT, Demarco FF, Goettems ML. Do maternal depression and anxiety influence children's oral health-related quality of life? Community Dent Oral Epidemiol. 2017 Oct;45(5):398-406. doi: 10.1111/cdoe.12303. Epub 2017 Apr 17. PMID 28417515
- [Background] Gavic L, Tadin A, Mihanovic I, Gorseta K, Cigic L. The role of parental anxiety, depression, and psychological stress level on the development of early-childhood caries in children. Int J Paediatr Dent. 2018 Nov;28(6):616-623. doi: 10.1111/ipd.12419. Epub 2018 Aug 24. PMID 30144198
- [Background] Burgette JM, Polk DE, Shah N, Malik A, Crout RJ, Mcneil DW, Foxman B, Weyant RJ, Marazita ML. Mother's Perceived Social Support and Children's Dental Caries in Northern Appalachia. Pediatr Dent. 2019 May 15;41(3):200-205. PMID 31171071
- [Background] Mohammad S, Almakran IW, Al-Montashri AS, Mursi AM, Alharbi SM, Pasha TS, Khalid I. Depression, anxiety and stress and their associated social determinants in the Saudi college students. Health Psychol Res. 2020 Dec 30;8(3):9263. doi: 10.4081/hpr.2020.9263. eCollection 2020 Dec 30. PMID 33553792